CLINICAL TRIAL: NCT03852615
Title: The Influence of Ovarian Torsion and Surgical De-torsion on Ovarian Reserve
Brief Title: Ovarian Reserve After Ovarian Torsion
Acronym: OTAMH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Aya Mohr-Sasson, Principal Investigator, Sheba Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 5646-18-SMC
Record Dates: First submitted 2019-02-12; First posted 2019-02-25 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Ovarian Torsion
Keywords: Ovarian Torsion; Laparoscopy; Anti Mullarian Hormone (AMH)
MeSH Terms: conditions — Ovarian Torsion

STUDY DESIGN:
Intervention Model Description: This is a prospective case control study including all women admitted to the gynecological emergency room with high clinical suspicious of ovarian torsion, that are planned to go through laparoscopic surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ovarian torsion (Experimental): Women admitted to the gynecological emergency room with high clinical suspicious of ovarian torsion, that went through laparoscopic ovarian de-torsion surgery
  Interventions: Diagnostic Test: Pre operation Blood sample for AMH; Diagnostic Test: 3 month post operation blood sample for AMH
- No ovarian torsion (Other): Control group - Women admitted to the gynecological emergency room with high clinical suspicious of ovarian torsion and went through laparoscopic surgery, however no ovarian torsion has been demonstrated
  Interventions: Diagnostic Test: Pre operation Blood sample for AMH; Diagnostic Test: 3 month post operation blood sample for AMH

INTERVENTIONS:
Diagnostic Test: Pre operation Blood sample for AMH — Blood sample for Anti Mullarian Hormone (AMH) analysis will be taken during preparation for surgery, while inserting vein line and taking the customary blood samples.
Diagnostic Test: 3 month post operation blood sample for AMH — Additional blood sampling that will include a single tube containing 3 cc of blood for analysis of AMH will be taken three month from operation.

SUMMARY:
Ovarian torsion is a relatively common gynecological emergency, usually presenting as acute lower abdominal pain. Due to patient's presentation diversity, the diagnosis is clinical and requires integration of different factors and the exclusion of other non-gynecological pathologies. Surgery is the definitive treatment and may still be effective after several hours of symptoms. Delay in treatment can impact fertility adversely. The aim of this study is to evaluate the change in anti mullarian hormone before and after laparoscopic de-torsion of the ovary in our medical center compared to controls.

DETAILED DESCRIPTION:
Ovarian torsion is a relatively common gynecological emergency, usually presenting as acute lower abdominal pain. The underlying pathophysiology involves torsion of the ovarian tissue on its pedicle leading to reduced venous return, stromal edema, internal hemorrhage and infarction with the subsequent sequelae.

The diagnosis of ovarian torsion is not an easy diagnosis to make and it is commonly missed. Signs and symptoms often mimic other disorders such as appendicitis, pyelonephritis, and nephrolithiasis. Abnormal arterial blood flow on ultrasound does not rule out ovarian torsion and not every patient will have a mass on imaging or a palpable mass on examination. Patients may have symptoms for several hours or days, and thus, may present even with a longer duration of symptoms. Due to patient's presentation diversity, the diagnosis is clinical and requires integration of different factors and the exclusion of other non-gynecological pathologies.

Surgery is the definitive treatment and may still be effective after several hours of symptoms. Delay in treatment can impact fertility adversely. Conservative laparoscopic surgery for de-torsion is considered a safe procedure to preserve ovarian function in women with adnexal torsion and is mostly salvaged ovaries will maintain viability after de-torsion.

Although the main reason for emergent operation is to rescue ovarian tissue in order to preserve future fertility, studies are scarce and mostly performed on animals models. Yasa et al, studied the ovarian reserve evaluated by antral follicle count and AMH levels in 11 patients with ovarian torsion that underwent laparoscopic de-torsion rand found no significant change in serum AMH level at 1 and 3 months after laparoscopic de-torsion compared with the preoperative levels, however sample size was small. The aim of this study is to evaluate the change in anti mullarian hormone before and after laparoscopic de-torsion of the ovary in our medical center compared to controls.

Material and methods This is a prospective case control study including all women admitted to the gynecological emergency room with high clinical suspicious of ovarian torsion, that are planned to go through laparoscopic surgery. Study group will include women that will be diagnosed with ovarian torsion during operation that will be compared to controls- women that ovarian torsion was not demonstrated.

All women will sign informed consent before admitted to operation room after given explanation from one of the study researchers. During preparation to surgery, while inserting vein line and taking the customary blood samples, additional tube that will include 3 cc of blood, will be taken for Anti Mullarian Hormone (AMH) analysis in the endocrinology laboratories. All women will be coordinated by the study coordinator for a second visit in the gynecological ward, three month from operation for additional blood sampling that will include a single tube containing 3 cc of blood for analysis of AMH.

ELIGIBILITY:
Inclusion Criteria:

* Suspected ovarian torsion
* Laparoscopy operation - explorative / de-torsion of ovary

Exclusion Criteria:

* Severe endometriosis
* Known premature ovarian failure
* Past ovarian operations other than de- torsion

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women
Enrollment: 81 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Anti Mullarian Hormone (AMH) change | From date of recruitment before laparoscopy until three month after laparoscopy
  The change in Anti Mullarian Hormone (AMH) levels before and three month after laparoscopy

SECONDARY OUTCOMES:
Ovarian change in color after de-torsion during laparoscopy | During laparoscopic operation, and through study completion, an average of 1 year
  Ovarian color before and after de-torsion , as described by the operator (black- necrotic , blue- highly congested, red- hyperemic , pink-normal)
Time to de-torsion | Estimated time from admission to the emergency room to de-torsion during laparoscopy in minutes
  Time from admission to the emergency room to de-torsion in minutes
Ovarian size after de-torsion during laparoscopy | During laparoscopic operation, and through study completion, an average of 1 year
  Estimated size of the ovary in centimeters

CONTACTS AND LOCATIONS:
Overall Officials: Aya Mohr Sasson, Principal Investigator — Sheba Medical Center, Tel-Hashomer
Locations (1):
- Aya Mohr Sasson, Ramat Gan, Please Select, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Asfour V, Varma R, Menon P. Clinical risk factors for ovarian torsion. J Obstet Gynaecol. 2015;35(7):721-5. doi: 10.3109/01443615.2015.1004524. Epub 2015 Jul 27. PMID 26212687
- [Result] Robertson JJ, Long B, Koyfman A. Myths in the Evaluation and Management of Ovarian Torsion. J Emerg Med. 2017 Apr;52(4):449-456. doi: 10.1016/j.jemermed.2016.11.012. Epub 2016 Dec 14. PMID 27988260
- [Result] Grunau GL, Harris A, Buckley J, Todd NJ. Diagnosis of Ovarian Torsion: Is It Time to Forget About Doppler? J Obstet Gynaecol Can. 2018 Jul;40(7):871-875. doi: 10.1016/j.jogc.2017.09.013. Epub 2018 Apr 19. PMID 29681508
- [Result] Fujishita A, Araki H, Yoshida S, Hamaguchi D, Nakayama D, Tsuda N, Khan KN. Outcome of conservative laparoscopic surgery for adnexal torsion through one-stage or two-stage operation. J Obstet Gynaecol Res. 2015 Mar;41(3):411-7. doi: 10.1111/jog.12534. Epub 2014 Nov 3. PMID 25363700
- [Result] Dasgupta R, Renaud E, Goldin AB, Baird R, Cameron DB, Arnold MA, Diefenbach KA, Gosain A, Grabowski J, Guner YS, Jancelewicz T, Kawaguchi A, Lal DR, Oyetunji TA, Ricca RL, Shelton J, Somme S, Williams RF, Downard CD. Ovarian torsion in pediatric and adolescent patients: A systematic review. J Pediatr Surg. 2018 Jul;53(7):1387-1391. doi: 10.1016/j.jpedsurg.2017.10.053. Epub 2017 Nov 16. PMID 29153467
- [Result] Kaya C, Turgut H, Cengiz H, Turan A, Ekin M, Yasar L. Effect of detorsion alone and in combination with enoxaparin therapy on ovarian reserve and serum antimullerian hormone levels in a rat ovarian torsion model. Fertil Steril. 2014 Sep;102(3):878-884.e1. doi: 10.1016/j.fertnstert.2014.06.007. Epub 2014 Jul 1. PMID 24996496
- [Result] Parlakgumus HA, Aka Bolat F, Bulgan Kilicdag E, Simsek E, Parlakgumus A. Atorvastatin for ovarian torsion: effects on follicle counts, AMH, and VEGF expression. Eur J Obstet Gynecol Reprod Biol. 2014 Apr;175:186-90. doi: 10.1016/j.ejogrb.2014.01.017. Epub 2014 Jan 20. PMID 24507756
- [Result] Yasa C, Dural O, Bastu E, Zorlu M, Demir O, Ugurlucan FG. Impact of laparoscopic ovarian detorsion on ovarian reserve. J Obstet Gynaecol Res. 2017 Feb;43(2):298-302. doi: 10.1111/jog.13195. Epub 2016 Dec 8. PMID 27928855